CLINICAL TRIAL: NCT03212599
Title: Quantitative Analysis of the Expression of Dementia-relevant Genes by Intake of the Drug Disulfiram
Brief Title: Disulfiram as a Modulator of Amyloid Precursor Protein-processing
Acronym: DIMAP
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, K. Lieb, Director, Johannes Gutenberg University Mainz
Other Study IDs: DIMAP
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Alcohol Addiction
Keywords: APP-processing; Disulfiram; ADAM10; Alzheimer's disease; blood
MeSH Terms: conditions — Alcoholism; Alzheimer Disease 10; Alzheimer Disease | interventions — Disulfiram

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples of each participant are retained and stored at -80.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Disulfiram — alcohol addicted patients receive an oral Disulfiram application as recrudescence prevention after successful detoxication
  Other Names: Antabus

SUMMARY:
A causal therapeutic approach for treatment of Alzheimer's disease has not been established so far. The protein ADAM10 represents a promising target for an A-beta peptide preventing strategy. Treatment of human neuronal cells with Disulfiram, a drug which is used in clinical routine for recrudescence prevention of alcohol dependency, revealed an increased expression of ADAM10. This finding indicates a neuroprotective potential of Disulfiram. The investigators' research purpose aims at the verification of the results obtained in cell culture experiments in the human organism. Therefore, include alcohol addicted patients were included, which take the drug Disulfiram for recrudescence prevention, in our study. Patients are recruited from the patient-collective of the University Medical Center Mainz and the Central Institute for Mental Health Mannheim. Blood samples (max. 5 ml) are taken from the participants before the intake of Disulfiram and about two weeks after treatment. Demographic data are collected (such as age or onset of addiction). Gene expression is analyzed via reverse transcription polymerase chain reaction(RT-PCR) from blood cell-derived messenger ribonucleic acid (mRNA).

ELIGIBILITY:
Inclusion Criteria:

ambulant or stationary patients, which receive Disulfiram for recrudescence prevention

Exclusion Criteria:

Diagnosed Alzheimer's dementia Previous Disulfiram treatment less than four weeks before baseline blood collection

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruited are alhohol addicted patients, which take Disulfiram as recrudescence prevention after successful detoxication. Patients between 20 and 60 years of age are included in the study independent from gender or ethnic background
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-05; Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
expression of ADAM10 | August 2016
  expression of ADAM10 in the collected blood samples measured by quantitation of the mRNA amount using RealTime-RT-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Endres, Principal Investigator — Medical Center Johannes Gutenberg University

IPD SHARING:
Plan to Share IPD: Yes
availability by publication
Time Frame: The data will be published in 2017/18. Availabilty will depend on the Chosen Journal.

REFERENCES:
- [Derived] Saifi MA, Shaikh AS, Kaki VR, Godugu C. Disulfiram prevents collagen crosslinking and inhibits renal fibrosis by inhibiting lysyl oxidase enzymes. J Cell Physiol. 2022 May;237(5):2516-2527. doi: 10.1002/jcp.30717. Epub 2022 Mar 13. PMID 35285015